CLINICAL TRIAL: NCT00278031
Title: Quality of Life in Children Cured of Retinoblastoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Israel Cancer Association (Other)
Responsible Party: Principal Investigator, Michael Weintraub, DIrector, Pediatric Hematology Oncology, Hadassah Medical Organization
Other Study IDs: qolrb-HMO-CTIL
Record Dates: First submitted 2006-01-17; First posted 2006-01-18 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Retinoblastoma
Keywords: Retinoblastoma; Quality of life
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to assess the quality of life of children who have been cured of retinoblastoma - a malignant eye tumor. The study is questionnaire-based, and uses standardized quality of life assessment tools.

DETAILED DESCRIPTION:
Retinoblastoma is the most common eye tumor of children. It can present in one eye (unilateral) or in both eyes (bilateral). The bilateral form is always hereditary.

Retinoblastoma is a highly curable tumor. Using a combination of surgery, chemotherapy, radiation and local treatment modalities to the eye, over 98% of patients are cured. This means that most children diagnosed with retinoblastoma will become long-term survivors.

The use of surgery (taking out one eye), chemotherapy, and radiation may be associated with long term side-effects, some of which may have significant impact on the quality of life of the child. In addition, in case where the disease is hereditary, additional psychological issues arise.

The aim of our study is to assess, in a comprehensive and standardized fashion, the long term quality of life in children who were treated for retinoblastoma, and who are currently alive and well.

The assessment will include the use of questionnaires that assess quality of life, as well as participation in age-appropriate activities.

Each child, and his/her parent, will be interviewed and the questionnaires completed. The process will take about one hour for each child. No risk or discomfort to the child is involved.

ELIGIBILITY:
Inclusion Criteria:

* Past treatment for retinoblastoma

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Long term survivors of childhood retinoblastoma
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2006-03; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change in quality of life | Baseline and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Weintraub, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Yes